CLINICAL TRIAL: NCT01713192
Title: Registry for Perioperative Data in Patients Undergoing Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Associate Professor, Seoul National University Hospital
Other Study IDs: YSJeon_Registry
Record Dates: First submitted 2012-10-22; First posted 2012-10-24 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Cardiac Surgical Procedures; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cardiac surgery

SUMMARY:
The purpose of this registry is to obtain perioperative data in patients undergoing cardiac surgery and find out relations between the data and investigate several causes affecting postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac surgery

Exclusion Criteria:

* refused to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
perioperative data | 1 year after surgery
  To obtain the perioperative data in patients undergoing cardiac surgery. Data will be collected including demographics, surgery and postoperative complications.
  In addition, laboratory data such as coagulation and cytokine will be obtained. Intraoperative monitoring including bispectral index, cerebral oximeter, tissue oxygen saturation [InspectraTM StO2 (Hutchinson Technology Inc., MN, USA)], cardiac index [FloTrac/EV1000 (Edwards Lifesciences, Irvine, CA, USA), VolumeView/EV1000 (Edwards Lifesciences, Irvine, CA, USA), Vigilance II (Edwards Lifesciences, Irvine, CA, USA)] and mixed venous oxygen saturation will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Cho YJ, Koo CH, Kim TK, Hong DM, Jeon Y. Comparison of cardiac output measures by transpulmonary thermodilution, pulse contour analysis, and pulmonary artery thermodilution during off-pump coronary artery bypass surgery: a subgroup analysis of the cardiovascular anaesthesia registry at a single tertiary centre. J Clin Monit Comput. 2016 Dec;30(6):771-782. doi: 10.1007/s10877-015-9784-6. Epub 2015 Oct 1. PMID 26429135
- [Derived] Kim TK, Cho YJ, Min JJ, Murkin JM, Bahk JH, Hong DM, Jeon Y. Microvascular reactivity and clinical outcomes in cardiac surgery. Crit Care. 2015 Sep 4;19(1):316. doi: 10.1186/s13054-015-1025-3. PMID 26337035